CLINICAL TRIAL: NCT01489943
Title: A Single Centre, Single Sequence, Open-Label, Repeat-Dose Study to Investigate the Effect of GSK1605786 on Hepatic Cytochrome P450, and BCRP and OATP1B1 Transport in Healthy Adult Subjects
Brief Title: A Study to Investigate the Effect of GSK1605786 on Hepatic Cytochrome P450, and BCRP and OATP1B1 Transport in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 114671
Record Dates: First submitted 2011-12-01; First posted 2011-12-12 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Midazolam; Pioglitazone; Omeprazole; Rosuvastatin Calcium

ARMS (1):
- All subjects receiving treatment (Experimental): During the treatment subjects will receive Midazolam 3 mg on Day 1, Pioglitazone 15 mg on Day 2, Omeprazole 40 mg on Day 3, Rosuvastatin 10 mg on Day 4, GSK1605786 500 mg twice daily (BID) from Day 5 to 10, GSK1605786 500 mg BID + Midazolam 3 mg on Day 11, GSK1605786 500 mg BID + Pioglitazone 15 mg on Day 12, GSK1605786 500 mg BID + Omeprazole 40 mg on Day 12, GSK1605786 500 mg BID + Rosuvastatin 10 mg on Day 14 as single sequence.
  Interventions: Drug: GSK1605786 500 mg; Drug: Midazolam 3 mg; Drug: Pioglitazone 15 mg; Drug: Omeprazole 40 mg; Drug: Rosuvastatin 10 mg

INTERVENTIONS:
Drug: GSK1605786 500 mg — Subjects will receive 500 milligram (mg) (2 doses of 250 mg) GSK1605786 hard gelatin capsules twice daily orally on Days 5 to 14. GSK1605786 will be administered with 240 milliliter (mL) of water.
Drug: Midazolam 3 mg — Subjects will receive 3 mg oral syrup of Midazolam once daily on Day 1 and Day 11. Midazolam will be administered with 240 mL of water.
Drug: Pioglitazone 15 mg — Subjects will receive 15 mg tablet of pioglitazone orally once daily on Day 2 and Day 12. Pioglitazone will be administered with 240 mL of water.
Drug: Omeprazole 40 mg — Subjects will receive 40 mg hard gelatin capsules of Omeprazole once daily on Days 3 and 13. Omeprazole will be administered with 240 mL of water.
Drug: Rosuvastatin 10 mg — Subjects will receive 10 mg tablet of Rosuvastatin orally once daily on Days 4 and 14. Rosuvastatin will be administered with 240 mL of water.

SUMMARY:
The purpose of this study is to test the effects of study drug (GSK1605786) on the blood levels of multiple commonly used drugs that are given to measure how your liver breaks down the study drug. These commonly-used drugs are midazolam, pioglitazone, omeprazole, and rosuvastatin which will determine the effect of GSK1605786 on how the body breaks down (metabolizes) these commonly-used drugs. Blood samples for pharmacokinetic analysis of GSK1605786, and two metabolites, [GSK2635622 (CCX062) and GSK2656694 (CCX304)] and four probe substrates will be collected over a 24-hour period after administration. Safety will be assessed by the measurement of vital signs, cardiac monitoring, collection of adverse event assessments and laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* Aspartate transaminase, alanine transaminase, alkaline phosphatase and bilirubin less than or equal to 1.5x the upper limit of normal (isolated bilirubin >1.5x the upper limit of normal is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if in the opinion of the Investigator the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of; non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<147 pmol/L) is confirmatory].
* Body weight more than or equal to 60 kg and BMI within the range 19 - 30 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form (including participation in pharmacogenetics research).
* QTc < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or Hepatitis B core antibody or positive Hepatitis C antibody result within 3 months of screening
* Current illness or disability that may affect the interpretation of clinical data, or otherwise contraindicates participation in this clinical study (e.g., an unstable cardiovascular, autoimmune, renal, hepatic, pulmonary, endocrine, metabolic, gastrointestinal, haematologic, or neurological condition or mental impairment)
* Current or pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic or renal function, that could interfere with the absorption, metabolism, or excretion of the study drugs; including but not limited to liver disease and known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 ml) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort [Hypericum perforatum], kava, ephedra [ma huang], gingko biloba, DHEA, vohimbe, saw palmetto, panaz ginseng, red yeast rice) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication and through the duration of the study, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety. Herbal medications include, but are not limited to: traditional Chinese, Korean and Japanese medicines, Panaz ginseng, Gingko biloba or St John's wort (Hypericum perforatum) or any Traditional Chinese herbal medicines (TCM) South Asian Ayurvedic medicine, Traditional Korean Medicines and Japanese Kampo.
* Use of aspirin, aspirin-containing compounds, salicylates or nonsteroidal anti-inflammatory drugs (NSAIDs) within 48 hours of the first dose and is unwilling to abstain from use of these medications until the last pharmacokinetic sample has been collected.
* Use of liquid antacids (e.g. Maalox, Mylanta, Amphogel, milk of magnesia) or tablets (including chewable) antacids (e.g. TUMS™) within 48 hours of the first dose and is unwilling to abstain from use of these medications until the last dose of study medication.
* Use of digoxin or related cardiac glycoside (e.g digitoxin, deslanoside, lanatoside C, metildigoxin) within 7 days prior to screening and throughout the study.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive serum hCG test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening. This includes chewing tobacco, Gutka, hand-rolled tobacco cigarettes, Biddis, cigars, and Snuff.
* Use of caffeine- or theobromine-containing beverages (e.g., coffee, tea, certain colas, green tea and oolong tea, Yerba Mate, Guarana, and South American cocoa) and foods (e.g., chocolate), or alcohol-containing beverages within 72 hours prior to dosing
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice, pummelos, exotic citrus fruits, grapefruit hybrids, fruit juice blends, apple or orange juice, vegetables from the mustard green family [e.g., kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, mustard] and charbroiled meats from 7 days prior to the first dose of study medication.
* Confirmed diagnosis of coeliac disease, those who follow a gluten-free diet to manage symptoms of suspected coeliac disease and subjects with a positive serologic test for tissue Transglutaminase, tTG (to screen for undiagnosed coeliac disease).
* Active or latent tuberculosis (TB) infection: All subjects will be tested with TB skin test (Mantoux test) and those with positive test result will be excluded.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-09-19 (Actual); Primary Completion 2011-11-10 (Actual); Study Completion 2011-11-10 (Actual)

PRIMARY OUTCOMES:
To investigate the potential of GSK1605786 to inhibit or induce drug metabolism via various CYP enzymes | 16 Days
  Midazolam AUC(0-infinity) following oral administration of midazolam alone (Day 1) and in combination with GSK1605786 (Day 11).Pioglitazone AUC(0-infinity) following oral administration of pioglitazone alone (Day 2) and in combination with GSK1605786 (Day 12).Omeprazole and 5-hydroxyomeprazole AUC(0-infinity) following oral administration of omeprazole alone (Day 3) and in combination with GSK1605786 (Day 13).
To investigate the potential of GSK1605786 to inhibit the BCRP and/or OATP1B1 transporters | 16 Days
  Rosuvastatin AUC(0-infinity) following oral administration of rosuvastatin alone (Day 4) and in combination with GSK1605786 (Day 14).

SECONDARY OUTCOMES:
To assess the safety and tolerablity of repeat oral doses of GSK1605786 | 21 Days
  Safety and tolerability during dosing with GSK1605786, alone and in combination with the various probe substrates. As assessed by adverse events, changes in vital signs, ECG, and hematology, clinical chemistry and urinalysis tests.
To determine the exposure of two metabolites, GSK2635622 (CCX062) and GSK2656694 (CCX304), relative to GSK1605786 (parent compound) following single and repeat administration of GSK1605786. | 16 Days
  Pharmacokinetic parameters [AUC(0-infinity), AUC(0-t), AUC(0-tau), Cmax, tmax, and half-life (t1/2)] of GSK1605786 after single and repeat administration of GSK1605786. Pharmacokinetic parameters [AUC(0-infinity), AUC(0-t), AUC(0-tau), Cmax, tmax, and half-life (t1/2)] of two metabolites of GSK1605786, GSK2635622 (CCX062) and GSK2656694 (CCX304) following single and repeat administration of GSK1605786.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States

REFERENCES:
- See also: Results for study 114671 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/114671?search=study&search_terms=114671#rs